CLINICAL TRIAL: NCT00577070
Title: Evaluation of the H-Coil Transcranial Magnetic Stimulation(TMS) Device- Augmentation for Drug Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Dr. Oded Rosenberg, Beer Yaakov MHC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TMS-204CTIL
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-01

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- H1 (Active Comparator): Includs 20 patients.These patients will be given 4 weeks (5 days a week) of deep TMS,20 minutes each session, to the left prefrontal cortex using H1 coil, in frequency of 20 HZ, with intensity of 120 % of motor threshold. H1-coil is an extracorporeal device positioned on the patient's scalp, designed to stimulate deep prefrontal brain regions, preferentially in the left hemisphere. The effective part of the coil, which has contact with the patient's scalp, includes 14 strips of 7-12 cm length. These strips are oriented in an anterior-posterior axis.This coil stimulates neuronal fibers in anterior-posterior orientation.
  During deep TMS exposure patients will listen to a clinical interview in which they describe the different expressions of their depression including their ruminations and depressive schemas.
  Interventions: Device: TMS
- H2 (Experimental): Includs 20 patients.These patients will be given 4 weeks (5 days a week) of deep TMS, 20 minutes each session, to the prefrontal cortex bilateraly using H2 coil, in frequency of 0.1 HZ, with intensity of 120 % of motor threshold. H2-coil is designed to stimulate deep prefrontal brain regions bilaterally (without any preferencefor either hemisphere). The effective part of the coil, which has contact with the patient's scalp, includes 10 strips of 14-22 cm length.These strips are oriented in a right-left direction (lateral-medial axis).This coil is destined to stimulate lateral-medial neuronal fibers. During deep TMS exposure patients will listen to a clinical interview in which they describe the different expressions of their depression including their ruminations and depressive schemas.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation (TMS) is a new tool in neuropsychiatry. This method is based on creating pre determined magnetic fields, which alternate rapidly. The magnetic fields are intended to cause electric induction in the brain cells and, as a consequence, generation of action potentials. The magnetic stimulation is delivered/ generated by a coil, positioned on the patient's scalp, inducing nerve stimulation within the brain. Therefore, when placed over the motor cortex, the magnetic stimulation creates Muscular Evoked potential, which can be measured by EMG.

SUMMARY:
There is a general consensus of efficacy of TMS in treatment of major depression,yet results are not satisfying.A new coil ("H"-coil, recently invented in Weizmann Institute of Science, Neurobiology Department, Rehovot, Israel) is supposed to be capable of stimulating deeper brain structures than conventional coils.TMS using this coil was named by its developers as "deep TMS" and will hence be refered to by this name.

So far, deep TMS have studied in Israel with promising sucssess in patients with Major depression (An on-going study).A safety study with good results have been recently published.The aim of this study is to reinforce initial results in major depression using deep TMS.

DETAILED DESCRIPTION:
A group of 40 patients with major depression will be randomly assigned to deep TMS with H-1 coil in frequency of 20 HZ or H-2 coil in frequency of 0.1 HZ with 120% of motor threshold to the prefrontal cortex . No change in anti-depressant medication one month prior to study is a prerequisite.Deep TMS will be administered for 4 weeks.During TMS exposure subjects will be exposed to a conversation in which they talk about their depression and their ruminations.Patients will be evaluated using Hamilton Depression Rating Scale (HAM-D24),Hamilton Anxiety Rating Scale (HAM-A),Clinical Global Impression - Improvement(CGI-I) ,Beck Depression Inventory (BDI),Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Right handed ,18-65 year old male or female subjects
* Diagnosed according to DSM-V-TR as suffering from Major depression using SCID interview
* Score of 22 or more in the Hamilton Depression Rating Scale (HAM-D24)
* The present depressive episode have been treated with at least 2 different anti-depressive drugs at peak doses for at least 6 weeks with not more than a partial response.Augmentation strategies may be included.

Exclusion Criteria:

Cardiac pacemaker implant, or a history of epilepsy, neurosurgery, or brain trauma patients suffering from chronic medical conditions of any sort:

* History of current hypertension
* History of seizure or heat convulsion
* History of epilepsy or seizure in first degree relatives
* History of head injury
* History of any metal in the head (outside the mouth)
* Known history of any metallic particles in the eye
* Implanted cardiac pacemaker or any intra-cardiac lines
* Implanted neuro-stimulators
* Surgical clips or any medical pumps
* History of frequent or severe headaches
* History of migraine
* History of hearing loss
* Known history of cochlear implants
* History of drug abuse or alcoholism
* Pregnancy or not using a reliable method of birth control (non-pregnancy will be proved by beta-HCG test)
* Systemic and metabolic disorders
* Inadequate communication skills or under custodial care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Treatment response defined as at least a 50% decrease in Hamilton Depression Rating Scale (HAM-D24). Remission is defined as below 8 in Hamilton Depression Rating Scale (HAM-D24) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Oded Rosenberg, M.D., Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer-Yaacov MHC, Beer Yaacov, Israel